CLINICAL TRIAL: NCT01485341
Title: Double Blind Randomized Placebo Controlled Multicenter Trial (Gluten vs Placebo) in Gluten Sensitive Subjects
Brief Title: Gluten Sensitivity in Non-Celiac Patients
Acronym: GS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Laura de Magistris, Senior Researcher, PhD, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 61-2-9-2011
Record Dates: First submitted 2011-11-17; First posted 2011-12-05 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Gluten Sensitivity
Keywords: gluten sensitivity
MeSH Terms: conditions — Celiac Disease | interventions — Glutens; substandard starch grain6 protein, rice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gluten (Active Comparator): gluten is administered blindly versus placebo for 15 days at 10 g/day
  Interventions: Dietary Supplement: gluten
- rice starch (Placebo Comparator): placebo (rice starch) will be administered blindly versus gluten for 15 days at 10 g/day
  Interventions: Dietary Supplement: rice starch

INTERVENTIONS:
Dietary Supplement: gluten — gluten is administered once a day at 10g/day for 15 days
  Arms: gluten
Dietary Supplement: rice starch — rice starch is administered once a day at 10 g/day for 15 days
  Arms: rice starch

SUMMARY:
The idea is to evaluate if the so called "Gluten Sensitivity" is a real clinical entity. Gluten sensitive (GS) persons are defined as those patients, being neither celiac or allergic to weat, who develop symptoms following gluten consumption. This will be achieved by evaluating a global symptom score in GS patients receiving gluten compared to those receiving placebo (primary end point). Symptoms to be evaluated: gastrointestinal (Gastrointestinal Symptom Rating Scale, GSRS); not-gastrointestinal (specifically built evaluation scale); VQV scale, built to evaluate quality of life. Gluten or placebo will be administered daily (10 g) for 15 days; for the 15 days before and 15 after all patients will stay on Gluten Free Diet (GFD). Besides clinical evaluation (each week for 6 weeks), intestinal permeability testing and blood sampling will be requested for the identification of possible markers (serological, gut barrier function, immunological and expression of tight junctions constitutive proteins) that may be of help to differentiate the condition of gluten sensitivity (GS) from that of Celiac Disease (CD)(secondary end point). Inclusion and exclusion criteria for patients enrolling are strictly dependant on the given "Gluten sensitivity" definition. We expect to experience a worsening of gastrointestinal and extra-gastrointestinal symptoms, from hours to days, with an increase in the overall symptom score, above the cut off, in at least 45% of GS subjects enrolled and that have received gluten compared to GS who received placebo.

DETAILED DESCRIPTION:
Gluten is the most important protein component of some grains, notably wheat, rye, and barley, which are the basis for a variety of flour and wheat derived alimentary products consumed throughout the world (bread, pasta, pizza etc). However the "engineering" of gluten-containing grains created the conditions for human diseases related to gluten exposure. These forms of gluten intolerance represent a heterogeneous set of conditions, including wheat allergy, Gluten Sensitivity and Celiac Disease, that, combined, affect about 10% of the general population. The frequency of not-celiac gluten intolerance is however still unknown, even though it is possible that these conditions have been undiagnosed and under-diagnosed by the physicians for long time. The state of immune responsiveness to wheat antigens, represents a complex process, and its establishment and maintenance are not completely elucidated. The most frequent diseases caused by wheat ingestion are T cell-mediated disorders, IgE-mediated allergic reactions and celiac disease (CD).

However, besides CD and wheat allergy, there are cases of gluten reactions in which neither allergic nor autoimmune mechanisms are involved. These are generally defined as gluten sensitivity (GS). Some individuals, who experience distress when eating gluten-containing products and show improvement when following a gluten-free diet, may have GS instead of CD. GS patients are unable to tolerate gluten and develop an adverse reaction when eating gluten that usually, and differently from CD, does not lead to small intestinal damage. While the gastrointestinal symptoms in GS may resemble those associated with CD, the overall clinical picture is generally less severe and is not accompanied by the concurrence of tTG autoantibodies or autoimmune disease. Typically the diagnosis is made by exclusion, and an elimination diet and "open challenge" (i.e., the monitored reintroduction of gluten-containing foods) are most often used to evaluate whether health improves with the elimination or reduction of gluten from the diet.

This has two major aims:

1. Evaluation of the effective dependence from the gluten of the clinical alterations presented by subjects with gluten sensitivity (GS). The study will be done after a period of gluten-free diet (washout of 15 days), comparing two groups of GS subjects: given gluten or placebo (15 days), followed by a further period (15 days) on gluten free diet .
2. identification of possible markers (serological, gut barrier function, immunological and expression of tight junctions constitutive proteins) that may be of help to differentiate, in humans, the condition of gluten sensitivity (GS) from that of Celiac Disease (CD); these markers might be of help in the early diagnosis of GS versus CD especially in the case of discordant serology.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age between 18-65 with signs/symptoms compatible with gluten-triggered disorders
* Patients testing negative for celiac disease either by biopsy Marsh 0-1 or those who are HLA-DQ2 and DQ8 negative, as well as tTG and EMA negative
* Patients that improved on a gluten free diet

Exclusion Criteria:

* Subjects diagnosed with celiac disease (positive TTG and/or EMA, and histology positive with Marsh II or above);
* Subjects diagnosed with wheat allergy
* Subjects with Type 1 Diabetes (T1D)
* Subjects with Inflammatory Bowel Disease (ulcerative colitis or Crohn's disease)
* Pregnancy
* Subjects with Helicobacter Pylori infection and other gastrointestinal infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Symptoms evaluation according to 3 scales: score after 2 weeks of gluten ingestion | Change from baseline at 2 weeks
  The evaluation will be made according to the score calculated on the basis of three evaluation scales: "Gastrointestinal Symptom Rating Scale "(GSRS), modified, provides a score ranging MIN=15/MAX=60; Extra-gastrointestinal symptoms evaluation scale, proposed on the basis of the symptoms most frequently observed in GS patients, provides a score ranging MIN=9/MAX=34; VQV scale proposed to evaluate the quality of life, provides a score ranging MIN=16/MAX=64. Total score can be no less than 37 (MIN) and not more than 146 (MAX), with a cut-off of 55.

SECONDARY OUTCOMES:
Bio-Markers to differentiate GS and CD | Change from baseline at 2 weeks
  The identification of possible markers (serological, gut barrier function, immunological and expression of tight junctions constitutive proteins) that may be of help to differentiate, in humans, the condition of gluten sensitivity (GS) from that of Celiac Disease (CD); these markers might be of help in the early diagnosis of GS versus CD especially when the serology is discordant.
Symptoms evaluation according to 3 scales: scores 2 weeks after completion of intervention | Return to baseline values at 4 weeks
  The evaluation will be made according to the score calculated on the basis of three evaluation scales: "Gastrointestinal Symptom Rating Scale "(GSRS), modified, provides a score ranging MIN=15/MAX=60; Extra-gastrointestinal symptoms evaluation scale, proposed on the basis of the symptoms most frequently observed in GS patients, provides a score ranging MIN=9/MAX=34; VQV scale proposed to evaluate the quality of life, provides a score ranging MIN=16/MAX=64. Total score can be no less than 37 (MIN) and not more than 146 (MAX), with a cut-off of 55.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sapone, MD, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (7):
- Center for Celiac Research & Treatment, Yawkey Center for Outpatients Care, Boston, Massachusetts, United States
- Italy (6):
  - Università Politecnica delle Marche, Ancona
  - Gastroenterologia ed Endoscopia digestiva, Ospedale San Giuseppe Moscati, Avellino
  - Gastroenterology, Second University of Naples, Naples
  - Internal Medicine, Policlinico di Palermo, Palermo
  - Gastroenterology, University of Salerno, Salerno
  - Ospedale "Casa Sollievo della Sofferenza" - IRCCS -, San Giovanni Rotondo (Foggia)